CLINICAL TRIAL: NCT02414503
Title: A Randomized, Placebo Controlled, Double-blind, 3-period Cross-over Study in Adult Patients With Autism Spectrum Disorders Evaluating Cognitive Response After Single- Dose Oxytocin 8 or 24 IU Intranasal Administration Using the OptiNose Bi-directional Nose-to-brain Device
Brief Title: Effects of Intranasal Administration of a Single Dose of Oxytocin Using a Novel Device in Adults With Autism Spectrum Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OptiNose AS (Industry)
Collaborators: Oslo University Hospital (Other); University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: SMR-2728; 2014-005452-26 (EudraCT Number)
Record Dates: First submitted 2015-03-31; First posted 2015-04-10 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Autism Spectrum Disorder
Keywords: oxytocin; social cognition
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 8IU intranasal oxytocin (Active Comparator): 8IU intranasal oxytocin delivered with the OptiNose Breath Powered Bi directional liquid device
  Interventions: Drug: 8IU intranasal oxytocin; Device: OptiNose Breath Powered Bi
- 24IU intranasal oxytocin (Active Comparator): 24IU intranasal oxytocin delivered with the OptiNose Breath Powered Bi directional liquid device
  Interventions: Drug: 24IU intranasal oxytocin; Device: OptiNose Breath Powered Bi
- Placebo (Placebo Comparator): Placebo delivered with the OptiNose Breath Powered Bi directional liquid device
  Interventions: Drug: Placebo; Device: OptiNose Breath Powered Bi

INTERVENTIONS:
Drug: 8IU intranasal oxytocin
  Arms: 8IU intranasal oxytocin
Drug: 24IU intranasal oxytocin
  Arms: 24IU intranasal oxytocin
Drug: Placebo
  Arms: Placebo
Device: OptiNose Breath Powered Bi

SUMMARY:
Oxytocin (OT) is a small, naturally occurring peptide currently in clinical use to stimulate lactation in breastfeeding women. The intranasal administration of OT has recently attracted attention as a potential novel treatment in several psychiatric disorders in autism. However, given the anatomy of the nasal cavity, the current design of nasal sprays would be expected to provide an inadequate delivery of medication to the areas of the nasal cavity where direct transport into the brain via the olfactory nerve could potentially occur. OptiNose has developed an intranasal delivery device that provides improved reproducibility of nasal delivery, improved deposition to the upper posterior regions of the nasal cavity where the olfactory nerve innervates the nasal cavity.

The primary objective of this study is to identify any differences between a single dose of 8 international units (IU) oxytocin, 24 IU oxytocin, and placebo delivered intranasally with the optimised OptiNose device in volunteers with Autism Spectrum Disorder. This will be measured in terms of performance on cognitive tests and physiological markers.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects between the ages of 18 and 35, both inclusive, with a confirmed diagnosis of autism spectrum disorder (ASD) diagnosis.
* Subjects must be in good general health, as determined by the investigator.
* Subject's pre-study physical examination, vital signs and electrocardiogram (ECG) must not show any clinically significant abnormalities as determined by the investigator.
* Subjects must be able to communicate well with the Investigator, to understand and comply with the requirements of the study, and to understand the oral and written patient information
* Provision of a signed, written informed consent.

Exclusion Criteria:

* Subjects showing major septal deviation or a significantly altered nasal epithelium.
* Subjects with evidence of previous nasal disease, surgery, and dependence on inhaled drugs.
* Subjects with current significant nasal congestion due to common colds.
* Subjects with a clinically relevant history of significant hepatic, renal, endocrine, cardiac, nervous, pulmonary, haematological or metabolic disorder.
* Psychiatric co-morbidity that requires intervention (e.g., psychosis spectrum disorders, suicide intent)
* Systemic illness requiring treatment within 2 weeks prior to Study Day 1.
* History of significant drug or alcohol abuse (as per WHO Alcohol use disorder identification test and drug use disorder identification test criteria) Subjects with a positive screen for alcohol or drugs of abuse at screening/admission will be excluded from participation in the study.
* Abnormal laboratory values which is deemed clinically significant by investigator.
* Full scale IQ < 75 (due to the prerequisite ability to complete self report measures).
* Known allergic reactions or hypersensitivity to any component of the study medication in the nasal spray, such as propyl parahydroxybenzoate (E216), methyl parahydroxybenzoate (E218) and chlorobutanol hemihydrate.
* Participation in any (other) clinical trial with an investigational medicinal product or medical device within 3 months prior to randomisation.
* Other unspecified reasons that, in the opinion of the investigator or the sponsor make the subject unsuitable for enrollment.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Performance on an emotion sensitivity test | 45 mins after oxytocin/placebo administration
  Participants will complete a task evaluating emotional expressions. These stimuli are identical to those published previously by Leknes et al., (2012).
Performance on a facial emotion morphing task | 45 mins after oxytocin/placebo administration
  Participants will complete a task evaluating faces that morph into different emotional expressions.

SECONDARY OUTCOMES:
Performance on the reading the mind in the eyes test | 45 mins after oxytocin/placebo administration
  Participants will complete the reading the mind in the eyes test
Performance on an emotional dot probe task | 45 mins after oxytocin/placebo administration
  Participants will complete an emotional dot probe task
Heart rate variability | 40 minutes after oxytocin/placebo administration
  Electrocardiogram data will be collected to assess heart rate variability, a measure of cardiac autonomic function.
Eyetracking | 45 mins after oxytocin/placebo administration
  An eyetracking device will measure eyegaze and pupillometry.

CONTACTS AND LOCATIONS:
Overall Officials: Ole A Andreassen, MD, PhD, Principal Investigator — University of Oslo
Locations (1):
- NORMENT, KG Jebsen Centre for Psychosis Research - TOP Study, Oslo, Norway

REFERENCES:
- [Background] Leknes S, Wessberg J, Ellingsen DM, Chelnokova O, Olausson H, Laeng B. Oxytocin enhances pupil dilation and sensitivity to 'hidden' emotional expressions. Soc Cogn Affect Neurosci. 2013 Oct;8(7):741-9. doi: 10.1093/scan/nss062. Epub 2012 May 29. PMID 22648957
- See also: Norwegian Centre for Mental Disorders Research — http://www.med.uio.no/norment/english/